CLINICAL TRIAL: NCT02484404
Title: Phase I/II Study of the Anti-Programmed Death Ligand-1 Antibody Durvalumab (MEDI4736) in Combination With Olaparib and/or Cediranib for Advanced Solid Tumors and Advanced or Recurrent Ovarian, Triple Negative Breast, Lung, Prostate and Colorectal Cancers
Brief Title: Phase I/II Study of the Anti-Programmed Death Ligand-1 Durvalumab Antibody (MEDI4736) in Combination With Olaparib and/or Cediranib for Advanced Solid Tumors and Advanced or Recurrent Ovarian, Triple Negative Breast, Lung, Prostate and Colorectal Can...
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 150145; 15-C-0145
Record Dates: First submitted 2015-06-25; First posted 2015-06-29 (Estimated); Last update posted 2025-11-25 (Actual); Status verified 2025-11-21

CONDITIONS: Colorectal Neoplasms; Breast Neoplasms
Keywords: Immune Checkpoint Inhibitor; PARP Inhibitor; VEGFR Inhibitor
MeSH Terms: conditions — Colorectal Neoplasms; Breast Neoplasms | interventions — olaparib; cediranib; durvalumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- P1 Durvalumab+C (Experimental): Ph I Durvalumab + cediranib dose escalation
  Interventions: Drug: Cediranib; Drug: Durvalumab
- P1 Durvalumab+O (Experimental): Ph I Durvalumab + olaparib dose escalation
  Interventions: Drug: Olaparib; Drug: Durvalumab
- P1 Durvalumab+O+C (Experimental): Ph I Durvalumab + olaparib + cediranib dose escalation
  Interventions: Drug: Olaparib; Drug: Cediranib; Drug: Durvalumab
- P2 Durvalumab+C (Experimental): Ph II Durvalumab + cediranib at RP2D
  Interventions: Drug: Cediranib; Drug: Durvalumab
- P2 Durvalumab+O (Experimental): Ph II Durvalumab + olaparib at RP2D
  Interventions: Drug: Olaparib; Drug: Durvalumab
- P2 Durvalumab+O+C (Experimental): Ph II Durvalumab + olaparib + cediranib at RP2D
  Interventions: Drug: Olaparib; Drug: Cediranib; Drug: Durvalumab

INTERVENTIONS:
Drug: Olaparib — Olaparib tablets will be given orally on a continuous dosing schedule. The DLT period will be one cycle, 28 days. MEDI4736 (3mg/kg or 10mg/kg IV) and Olaparib tablets (200 mg or 300 mg BID) Ph II - MEDI4736 + Olaparib at RP2D
  Arms: P1 Durvalumab+O; P1 Durvalumab+O+C; P2 Durvalumab+O; P2 Durvalumab+O+C
Drug: Cediranib — Cediranib will be given orally on a continuous dosing schedule. The DLT period will be one cycle, 28 days. MEDI4736 (10mg/kg IV) and Cediranib (15 mg or 20 mg or 30 mg daily) Ph II - MEDI4736 + Cediranib at RP2D
  Arms: P1 Durvalumab+C; P1 Durvalumab+O+C; P2 Durvalumab+C; P2 Durvalumab+O+C
Drug: Durvalumab — Ph I - Durvalumab will be administered once every 2 weeks for 12 months.

SUMMARY:
Background:

- Durvalumab is a drug that may help people s immune systems respond to and kill cancer cells. Olaparib is a drug that may inhibit repairing DNA damage of cancer cells. Cediranib is a drug that may stop the blood vessel growth of cancer cells. This study has two components. In the phase 1 component of the study, researchers want to investigate how well participants tolerate the combination of these drugs in treating advanced solid tumors, and in the phase 2 part of this study, researchers want to study if the combination treatments are effective in ovarian cancer.

Objectives:

- Phase 2 part of the study: To determine how effective this combination is in treating ovarian cancer.

Eligibility:

- Phase 2 part of the study: Adults age 18 or older with advanced or recurrent ovarian cancer that has no standard treatment.

Design:

* Participants will be screened with medical history, physical exam, and blood and urine tests. They will have CT or MRI scans. For these, they will lie in a machine that takes pictures of their bodies.
* Phase 2 part of the study requests the participants to have tumor samples removed.
* Participants will get Durvalumab through an IV. A small plastic tube will be inserted into a vein. The drug will be given every 4 weeks until disease progression.
* Participants will take olaparib or cediranib by mouth every day.
* Every 28 days will be 1 cycle. For cycle 1, participants will have 2 study visits. All other cycles, they will have 1 visit. At these visits, they will repeat the screening procedures.
* Patients will keep a drug and diarrhea diary.
* Patients on cediranib will monitor their blood pressure and keep a blood pressure diary.
* Participants who can become pregnant, or have a partner who can become pregnant, must practice an effective form of birth control.
* After 12 cycles, participants will have 1-3 months of follow-up.

DETAILED DESCRIPTION:
Background:

Disruption of the immune checkpoint PD-1/PD-L1 pathway yielded clinical activity in subsets of advanced solid tumors, such as melanoma and lung cancer.

Olaparib (O), a PARP inhibitor (PARPi), has demonstrated single agent activity in recurrent ovarian cancer (OvCa), and subsets of prostate, triple negative breast or lung cancers.

Our recent randomized phase 2 study showed that O and cediranib (C), a VEGFR1-3 inhibitor was clinically superior to O alone in platinum-sensitive recurrent OvCa.

We hypothesize that increased DNA damage by PARP inhibition and/or reduced angiogenesis by VEGFR inhibition will complement the anti-tumor activity of an immune checkpoint inhibitor, Durvalumab, in recurrent OvCa and other solid tumors.

Objectives:

Phase I: To determine the recommended phase II dose (RP2D) and the safety of doublet therapies (Durvalumab/olaparib [Durvalumab+O] and Durvalumab/cediranib [Durvalumab+C]) and triplet therapy (Durvalumab+O+C) in patients with advanced solid tumors.

Phase II Cohort 2 non-small cell lung cancer (NSCLC); Durvalumab+O and Durvalumab+C arms: To determine clinical efficacy as measured by progression-free survival (PFS)

Phase II Cohort 3 small cell lung cancer (SCLC); Durvalumab+O arm: To determine clinical efficacy as measured by ORR

Phase II Cohort 4 metasttaic castrate-resistant prostate cancer (mCRPC); Durvalumab+O arm: To determine clinical efficacy as measured by PFS

Phase II Cohort 5 triple negative breast cancer (TNBC); Durvalumab+O arm: To determine clinical efficacy as measured by ORR

Phase II Cohort 1 OvCa; Durvalumab+O, Durvalumab+C and Durvalumab+O+C arms: To determine clinical efficacy as measured by overall response rate (ORR)

Phase II Cohort 6 colorectal cancer (CRC): C+Durvalumab arm: To determine clinical efficacy as measured by PFS

Eligibility:

Phase I: Advanced or recurrent solid tumors with evaluable disease.

Phase II Cohort 1 Durvalumab+O, Durvalumab+C and Durvalumab+O+C arms: Advanced or recurrent OvCa

Phase II Cohort 2 Durvalumab+O and Durvalumab+C arms: Advanced or recurrent NSCLC

Phase II Cohort 3 Durvalumab+O arm: Advanced or recurrent SCLC

Phase II Cohort 4 Durvalumab+O arm: mCRPC

Phase II Cohort 5 Durvalumab+O arm: Advanced or recurrent TNBC

Phase II Cohort 6 C+Durvalumab arm: Advanced or recurrent CRC

Patients must be off prior chemotherapy, radiation therapy or biologic therapy for at least 3 weeks. mCPRC patients (Cohort 4) may be on hormonal therapy with GnRH agonists/antagonists.

Adults with ECOG performance status 0-2, and adequate organ and marrow function.

Design:

Phase I: Durvalumab+O, Durvalumab+C and Durvalumab+O+C will dose escalate simultaneously. Durvalumab will be administered once every 2 weeks or once every 4 weeks until disease progression. O tablets and C will be given orally on a continuous or intermittent dosing schedule. The DLT period will be one cycle, 28 days. Patients on the 2-week schedule greater than one year will be changed to the 4-week schedule until progression.

Durvalumab+O: Durvalumab (3 mg/kg or 10 mg/kg IV every 2 weeks, or a fixed dose of 1500 mg every 4 weeks) and O tablets (150 mg or 200 mg or 300 mg BID)

Durvalumab+C: Durvalumab (3 mg/kg or 10 mg/kg IV every 2 weeks, or a fixed dose of 1500 mg every 4 weeks) and C (15 mg or 20 mg or 30 mg daily or 5 days/week)

Durvalumab+O+C: Durvalumab (a fixed dose of 1500mg every 4 weeks) with O tablets (200 mg or 300 mg BID) and C (15 mg or 20 mg 5 days/week)

Phase II Cohort 1 OvCa Durvalumab+O arm: Patients will be treated with Durvalumab+O at RP2D (O 300mg tablets bid daily and Durvalumab at 1500 mg IV every 4 weeks).

Phase II Cohort 1 OvCa Durvalumab+C arm: Patients will be treated with Durvalumab+C at RP2D (C 20mg once a day [5 days on/2 days off] and Durvalumab at 1500 mg every 4 weeks).

Phase II Cohort 1 OvCa Durvalumab+O+C arm: Patients with OvCa (Cohort 1) will be treated with RP2D (O tablets 300mg BID, C 20mg once a day [5 days on/2 days off] and Durvalumab at 1500 mg every 4 weeks).

Phase II Cohort 2 NSCLC; Durvalumab+O arm: Patients will be treated with Durvalumab+O at RP2D (O 300mg tablets bid daily and Durvalumab at 1500 mg IV every 4 weeks).

Phase II Cohort 2 NSCLC; Durvalumab+C arm: Patients will be treated with Durvalumab+C at RP2D (C 20mg once a day [5 days on/2 days off] and Durvalumab at 1500 mg every 4 weeks).

Phase II Cohort 3 SCLC; Durvalumab+O arm: Patients will be treated with Durvalumab+O at RP2D (O 300mg tablets bid daily and Durvalumab at 1500 mg IV every 4 weeks).

Phase II Cohort 4 mCRPC; Durvalumab+O arm: Patients will be treated with Durvalumab+O at RP2D (O 300mg tablets bid daily and Durvalumab at 1500 mg IV every 4 weeks).

Phase II Cohort 5 TNBC; Durvalumab+O arm: Patients will be treated with Durvalumab+O at RP2D (O 300mg tablets bid daily and Durvalumab at 1500 mg IV every 4 weeks).

Phase II Cohort 6 CRC; C+Durvalumab arm: Patients in the Cohort 6 will be treated with C 20mg daily alone for 14 days followed by the combination at RP2D (C 20mg once a day [5 days on/2 days off] and Durvalumab at 1500 mg every 4 weeks).

Phase II Correlative studies: Research samples including whole blood, CTCs, cell free DNA and plasma will be obtained at pretreatment, prior to cycle 1 day 15, prior to cycle 3 day 1 and at progression. Mandatory baseline core biopsy and two optional biopsies will be obtained.

Patients will be evaluated for toxicity every 4 weeks by CTCAEv4.0, and for response every two cycles (8 weeks) by RECIST 1.1. Patients with mCRPC (Durvalumab+O Cohort 4) will be evaluated for response initially at 8 weeks then every 12 weeks using RECIST v1.1 criteria as per the Prostate Cancer Clinical Trials Working Group 2 (PCWG2).

ELIGIBILITY:
* ELIGIBILITY:

INCLUSION CRITERIA GENERAL:

* Patients must be at least 18 years of age.
* Patients must have adequately controlled blood pressure on a maximum of three antihypertensive medications.
* Patients who have the following clinical conditions are considered to be at increased risk for cardiac toxicities.

Patients with any cardiac history of the following conditions within 1 year prior to study enrollment are excluded from the study:

* Prior events including myocardial infarction, pericardial effusion, and myocarditis.
* Prior cardiac arrhythmia including atrial fibrillation and atrial flutter, or requiring concurrent use of drugs or biologics with pro-arrhythmic potential.
* NYHA Class II or greater heart failure.
* If cardiac function assessment is clinically indicated or performed, an LVEF less than normal per institutional guidelines, or <55%, if threshold for normal is not otherwise specified by institutional guidelines.
* QTc prolongation >470 msec or other significant ECG abnormality noted within 14 days of treatment.
* Hypertensive crisis or hypertensive encephalopathy.
* Clinically significant peripheral vascular disease or vascular disease, including rapidly growing aortic aneurysm or abdominal aortic aneurysm >5 cm or aortic dissection.
* Unstable angina.

  * Eligibility for patients with asymptomatic and a previous diagnosis of immune or inflammatory colitis, or patients with chronic diarrhea > 1 month without immune or inflammatory colitis is a PI decision on an individual patient basis.
  * Patients with a history of cerebrovascular accident or transient ischemic attack within 1 year prior to study enrollment are not eligible.
  * Patients with a history of previous clinical diagnosis of tuberculosis are not eligible.
  * Patients with a history of auto-immune disease requiring steroid maintenance, or history of primary immunodeficiency are not eligible.
  * HIV-positive patients on antiretroviral therapy are ineligible because of potential pharmacokinetic interactions with study drugs, however, patients with long-standing (>5 years) HIV on antiretroviral therapy > 1 month (undetectable HIV viral load and CD4 count > 150 cells/microL) may be eligible if the PI determines no anticipated clinically significant drug-drug interactions.
  * HBV-or HCV-positive patients are ineligible because of potential reactivation of hepatitis virus following steroids.
  * Patients with a history of allergic reactions attributed to compounds of similar chemical or biologic composition to MEDI4736, olaparib, cediranib, or to other humanized monoclonal antibodies, or a history of anaphylaxis, angioedema, laryngeal edema, serum sickness, or uncontrolled asthma, are not eligible.
  * Patients who have had prior immune checkpoint inhibitors, such as MEDI4736 or other PD1 or PD-L1 inhibitors or an anti-CTLA4 therapy are eligible.
  * Pregnant and breastfeeding women are excluded from this study.
  * Patients with any other concomitant or prior invasive malignancies are ineligible.

PHASE II MEDI4736 PLUS OLAPARIB OR CEDIRANIB STUDY ELIGIBILITY CRITERIA - OVARIAN CANCER

* Patients must have histologically or cytologically confirmed persistent or recurrent ovarian, fallopian tube, or primary peritoneal cancer and have received at least two prior regimens or who are platinum resistant or refractory during or after a first platinum containing regimen.
* Patients must have at least one lesion deemed safe to biopsy and be willing to undergo a mandatory baseline biopsy.
* Patients are allowed to have received prior PARPi, and/or anti-angiogenesis therapy including but not limited to thalidomide, bevacizumab, sunitinib, sorafenib, or other anti-angiogenics. However, patients who were treated with both olaparib and cediranib, either in combination or sequentially are not eligible. For this study, BSI-201 (iniparib) is not considered as PARPi.

PHASE II STUDY MEDI4736 PLUS OLAPARIB ELIGIBILITY CRITERIA TRIPLE NEGATIVE BREAST CANCER

* Patients must have histologically confirmed persistent or recurrent triple-negative breast cancer (TNBC)
* ER/PR/HER2 status needs to be documented either by an outside source or at NCI.
* Documentation of germline BRCA1 and BRCA2 mutation (gBRCAm) status will be required for eligibility.
* Patients must have measurable disease as defined by RECIST v1.1.
* Patients must have at least one lesion deemed safe to biopsy and be willing to undergo a mandatory baseline biopsy.
* Patients who have received prior PARPi are ineligible.
* Patients must not have evidence of CNS metastasis or leptomeningeal disease within one year prior to enrollment.

PHASE II MEDI4736 PLUS OLAPARIB OR CEDIRANIB STUDY ELIGIBILITY CRITERIA - NON-SMALL CELL LUNG CANCER

* Histologically or cytologically confirmed advanced NSCLC with at least one prior line of platinum-based chemotherapy (or treatment with EGFR, ALK, or BRAF-targeted tyrosine kinase inhibitors if tumors harbor an EGFR-sensitizing mutation, ALK translocation, or BRAF V600E mutation, respectively).
* Patients must have measurable disease as defined by RECIST v1.1.
* Patients must have at least one lesion deemed safe to biopsy and be willing to undergo a mandatory baseline biopsy.
* Patients who have received anti-angiogenesis therapy are eligible, including but not limited to thalidomide, bevacizumab, sunitinib, sorafenib, or other anti-angiogenics. However, patients who were treated with cediranib, either in combination or monotherapy are not eligible.
* Current or prior use of immunosuppressive medication within 28 days before the first dose of MEDI4736, with the exception of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone or an equivalent corticosteroid.
* Patients who have had prior PARPi are not eligible.
* Patients with prior history of pneumonitis and/or interstitial lung disease will be excluded.

PHASE II MEDI4736 PLUS OLAPARIB STUDY ELIGIBILITY CRITERIA - METASTATIC CASTRATE-RESISTANT PROSTATE CANCER

* Patients must have metastatic, progressive, castrate resistant prostate cancer (mCRPC).
* All patients must have at least one lesion deemed safe to biopsy and be willing to undergo a mandatory baseline biopsy.
* Patients must have received prior treatment with enzalutamide and/or abiraterone with the exception of patients who were treated with docetaxel and androgen deprivation therapy for metastatic castrate-sensitive prostate cancer and progressed on docetaxel treatment or who progress within one month of the last docetaxel dose.
* Patients must have undergone bilateral surgical castration or must agree to continue on GnRH agonists/antagonists for the duration of the study.
* Patients who have had progression of prostate cancer on prior docetaxel treatment for castrate sensitive disease are ineligible.
* Patients who have had prior treatment with PARPi are not eligible.
* Patients who have received radionuclide treatment within 6 weeks prior to the first dose of the study treatment are not eligible.
* Patients with any other concomitant or prior invasive malignancies are ineligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Actual)
Dates: Start 2015-06-29 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Ph II Determine overall response rate of Durvalumab-O and Durvalumab-C in patients with recurrent ovarian cancer | every 4 wks for toxicity and every 8 wks for response
  Overall response rate
Ph I Determine the recommended phase II dose (RP2D) and the safety of doublet therapies of Durvalumab/olaparib (Durvalumab-O) and Durvalumab/cediranib (Durvalumab-C) in patients with advanced solid tumors | 28 days
  Determination of the recommended phase II dose (RP2D) Safety: number of Adverse events

SECONDARY OUTCOMES:
Ph II Cohort 5 TNBC; Durvalumab+O arm: To determine PFS, safety by CTCAE v4.0, and potential relationship between pretreatment tumor PD-L1 expression obtained from biopsies and clinical response | every 28 days, every 8 weeks
  ORR + safety (adverse events)
Ph II Cohort 4 mCRPC; Durvalumab+O arm: To determine ORR, safety by CTCAE v4.0, duration of response and PSA responses. | every 28 days, every 8 weeks
  ORR + safety (adverse events), duration of response and PSA responses.
Ph II Cohort 3 SCLC; Durvalumab+O arm: To determine PFS and safety by CTCAE v4.0 | every 28 days, every 8 weeks
  PFS + Safety(adverse events)
Ph II Cohort 2 NSCLC; Durvalumab+O and Durvalumab+C arms: To determine ORR, and safety by CTCAE v4.0 | every 28 days, every 8 weeks
  ORR + Safety (adverse events)
Ph II Cohort 1 OvCa; Durvalumab+O, Durvalumab+C and Durvalumab+O+C arms: To evaluate PFS, safety by CTCAE v4.0, and potential relationship between pretreatment tumor PD-L1 expression obtained from biopsies and clinical response | every 28 days, every 8 weeks
  Progression-Free Survival (PFS) + Safety (adverse events) + PD-L1 expression obtained from biopsies and clinical response
Ph I of triplet tx:explore changes in peripheral immune subsets, plasma cytokines and circulating endothelial cells with safety and/or clinical outcome of Durvalumab+O+C | every 28 days
  Correlative laboratory research results + safety (adverse events) and/or clinical outcome
Ph I of triplet tx:determine the safety of Durvalumab+O+C | every 28 days
  Safety (adverse events)
Ph I of triplet tx:determine the potential relationship between PD-L1 expression obtained from archival tissue samples and clinical response | every 28 days
  PD-L1 expression obtained from archival tissue samples and clinical response
Ph I of triplet tx:determine the pharmacokinetics of the triplet and correlate with safety. | Cycle 1 Days 1 and 15; Cycles 2 and beyond Day 1
  Pharmacokinetics + Safety: adverse events
Ph I of triplet tx::determine preliminary response rates of Durvalumab+O+C using RECIST v1.1 | every 8 weeks
  Response: Preliminary response rate
Ph I doublet:determine the potential relationship between PD-L1 expression obtained from archival tissue samples and clinical response | every 28 days
  PD-L1 expression obtained from archival tissue samples and clinical response
Ph I doublet tx:determine preliminary response rates of the doublets using RECIST v1.1 | every 8 wks
  Response: Preliminary response rate
Ph I doublet tx: explore changes in peripheral immune subsets, plasma cytokines and circulating endothelial cells with safety and/or clinical outcome of Durvalumab+C | every 28 days
  Correlative laboratory research results + safety (adverse events) and/or clinical outcome
Ph I doublet tx: determine the safety of the doublets, Durvalumab+O and Durvalumab+C | every 28 days
  Safety: number of Adverse events
Ph I doublet tx: determine the pharmacokinetics of the doublets and correlate with safety. | Cycle 1 Days 1 and 15; Cycles 2 and beyond Day 1
  Pharmacokinetics + Safety: adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Takeo Fujii, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. @@@@@@In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.@@@@@@Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI. @@@@@@Genomic data are made available via dbGaP through requests to the data custodians.

REFERENCES:
- [Derived] Fujii T, Cimino-Mathews A, Lipkowitz S, Lee MJ, Nair J, Solarz BB, Zimmer A, Redd B, Levy EB, Rastogi S, Sato N, McCoy A, Steinberg SM, Lee JM. A Phase II Pilot Study of Anti-PD-L1, Durvalumab, and a PARP Inhibitor, Olaparib in Patients With Metastatic Triple-Negative Breast Cancer With or Without Germline BRCA Mutation. Cancer Med. 2025 Dec;14(23):e71220. doi: 10.1002/cam4.71220. PMID 41360639
- [Derived] Zimmer AS, Nichols E, Cimino-Mathews A, Peer C, Cao L, Lee MJ, Kohn EC, Annunziata CM, Lipkowitz S, Trepel JB, Sharma R, Mikkilineni L, Gatti-Mays M, Figg WD, Houston ND, Lee JM. A phase I study of the PD-L1 inhibitor, durvalumab, in combination with a PARP inhibitor, olaparib, and a VEGFR1-3 inhibitor, cediranib, in recurrent women's cancers with biomarker analyses. J Immunother Cancer. 2019 Jul 25;7(1):197. doi: 10.1186/s40425-019-0680-3. PMID 31345267
- [Derived] Karzai F, VanderWeele D, Madan RA, Owens H, Cordes LM, Hankin A, Couvillon A, Nichols E, Bilusic M, Beshiri ML, Kelly K, Krishnasamy V, Lee S, Lee MJ, Yuno A, Trepel JB, Merino MJ, Dittamore R, Marte J, Donahue RN, Schlom J, Killian KJ, Meltzer PS, Steinberg SM, Gulley JL, Lee JM, Dahut WL. Activity of durvalumab plus olaparib in metastatic castration-resistant prostate cancer in men with and without DNA damage repair mutations. J Immunother Cancer. 2018 Dec 4;6(1):141. doi: 10.1186/s40425-018-0463-2. PMID 30514390
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2015-C-0145.html